CLINICAL TRIAL: NCT03294486
Title: Safety and Efficacy of the ONCOlytic VIRus Armed for Local Chemotherapy, TG6002/5-FC, in Recurrent Glioblastoma Patients
Acronym: ONCOVIRAC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Transgene (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P150936; 2015-004452-21 (EudraCT Number)
Record Dates: First submitted 2017-08-02; First posted 2017-09-27 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Glioblastoma; Brain Cancer
Keywords: Glioblastoma; Oncolytic viruses
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Flucytosine

STUDY DESIGN:
Intervention Model Description: Phase 1 :
  Dose-escalation trial using an accelerated titration 3+3 design. Eligible patients will first be consecutively enrolled in a one-patient cohort at lowest dose level and then in 3-patients cohorts up to a DLT observation. All patients within a given cohort will be treated with the same dose schedule of TG6002. Following the 1st and 2nd infusion of TG6002 patients will be given oral 5-FC for 3 days starting on Day 5 and 12 and ending on Day 7 and 14, respectively. Following the 3rd infusion of TG6002 on Day 15, patients will be given oral 5-FC for 21 days starting on Day 19 and ending on Day 39 (end of treatment).
  Phase 2a Patients will be treated IV at the Recommended Phase 2 dose (RP2D).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of TG6002 and flucytosine (5-FC, Ancotil®) (Experimental): All patients within a given cohort will be treated with the same dose schedule of TG6002, administred as 3 weekly IV infusions at days 1, 8 and 15. following the 1st and 2nd infusions of TG6002, patients will be given oral 5-FC for 3 days starting on day 5 and 12 . following the 3rd infusion, patients will be given oral 5-FC for 21 days starting on day 19.
  Interventions: Drug: Combination of TG6002 and 5-flucytosine (5-FC, Ancotil®)

INTERVENTIONS:
Drug: Combination of TG6002 and 5-flucytosine (5-FC, Ancotil®) — Phase 1, TG6002 administered in a total volume of 250mL of saline solution (0.9 %) as three intravenous infusions at the following doses:
  * Dose 1 : 5.0 log10 pfu •Dose 2 : 6.0 log10 pfu •Dose 3 : 7.0 log10 pfu •Dose 4 : 7.5 log10 pfu
  * Dose 5 : 8.0 log10 pfu •Dose 6 : 8.5 log10 pfu Additional dose levels •Dose 2-1 : 5.5 log10 pfu •Dose 3-2 : 6.5 log10 pfu Phase 2a, treatment IV at the recommended Phase 2 dose 5-Flucytosine (5-FC) is provided in its commercial packaging with brand name ANCOTIL 500 mg, tablet (Ancotil®) marketed by MEDA Pharma: polypropylene tube containing 100 tablets.
    5-FC administered orally as 500 mg tablets taken 4 times per day (qid). Daily starting dose is 200 mg/kg. The daily dose will be adjusted at Day 19 following the measurement of 5-FC plasma concentration at steady state (Day 7), which should be kept below 100 mg/L.

SUMMARY:
Glioblastoma is the most common and the most aggressive primary brain cancer in adults. Indeed, despite very intensive treatments (i.e. maximal safe surgery, radiotherapy and several lines of cytotoxic chemotherapies), inducing significant adverse events, the prognosis of glioblastoma patients remains dismal with a median overall survival of ~15 months. Therefore, more efficient and less toxic therapies are urgently needed to improve survival and quality of life of glioblastoma patients.

The oncolytic virus TG6002 has shown efficacy and good safety profile in several preclinical models of glioblastoma in vitro (i.e. cell line) and in vivo (i.e. xenografts in Swiss/Nude mice). Comprehensive toxicology studies of TG6002/Flucytosine have been completed in rabbits and monkeys supporting safety investigations of TG6002/Flucytosine in human patients.

Taken these data all together, TG6002/Flucytosine appears as a very promising therapeutic strategy in glioblastoma patients that merits consideration for early phase clinical trial.

DETAILED DESCRIPTION:
Phase 1:

This is a Phase 1, open-label, dose-escalation trial using an accelerated titration 3+3 design in patients with recurrent glioblastoma. Eligible patients will first be consecutively enrolled in a one-patient cohort at lowest dose level and then in 3-patients cohorts up to a DLT observation. In case a DLT is observed specific rules apply to enrol additional (from 3 to 5) patients in the same cohort and to proceed to higher doses. All patients within a given cohort will be treated with the same dose schedule of TG6002, administered as 3 weekly IV infusions at Days 1, 8, and 15. Following the 1st and 2nd infusion of TG6002 on Day 1 and 8, patients will be given oral 5-FC for 3 days starting on Day 5 and 12 and ending on Day 7 and 14, respectively. Following the 3rd infusion of TG6002 on Day 15, patients will be given oral 5-FC for 21 days starting on Day 19 and ending on Day 39 (end of treatment). Patients will be followed until documented tumor progression.

The starting dose of 1 x 105 pfu is determined after toxicology results in the most sensitive species on which a security factor (100x) has been applied; accelerated titration will consist in one patient being administered with the starting dose and one-log dose increment between the three first cohorts.

The maximum tolerated dose (MTD) is defined as the highest TG6002 dose level at which at most 1 Dose-Limiting Toxicity (DLT) is observed in 6 patients exposed to that dose level.. The DLT period is defined as the interval between the first TG6002 IV infusion (Day 1) and the 8th day of the 21-day 5-FC treatment occurring on Day 26.

Between consecutive cohorts during dose escalation, an at least 3-week safety interval will be applied, starting from the completion of the DLT period of the last patient of the previous cohort (D26), before the infusion of the first patient of the next higher dose cohort (D47). The initiation of the next higher dose cohort will be determined following an analysis by the DSMB of the safety results from one cycle of TG6002 treatment in combination with 5-FC.

Phase 2a:

Based on the outcome of the Phase 1 dose-escalation cohorts, i.e. RP2D, the Phase 2a will include 24 patients. Patients will be treated IV at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Karnofsky performance status ≥ 70.
3. Histologically confirmed primary glioblastoma with unequivocal progression after at least the first line standard of care (concurrent chemoradiotherapy and adjuvant chemotherapy) at least 3 months after the completion of radiotherapy.
4. At least one measurable lesion, according to RANO criteria.
5. Availability of biological material (tumor) for review processes.
6. No treatment with another investigational drug within 4 weeks before inclusion.
7. No surgery within 4 weeks before inclusion.
8. If reoperation is conducted an early post-surgery MRI, within 48 hours is needed.
9. Standard-of-Care MRI showing a target lesion performed within 2 weeks prior to inclusion.
10. Stable or decreasing dosage of steroids for 7 days prior to the baseline MRI scan.
11. Non-enzyme inducing antiepileptic drugs (non-EIAED). Patients previously on EIAED must be switched to non-EIAED at least 2 weeks prior to inclusion.
12. No previous cancer except: (i) cancer in remission for at least 5 years, (ii) skin carcinoma, or (iii) in situ carcinoma of the uterine cervix.
13. Absence of any unstable disease (heart, liver, renal and respiratory failure).
14. Absence of serious conditions (as judged by the investigator) that could interfere with the treatment (i.e. infection, immunosuppression defined as CD4+ lymphocytes < 200/µL).
15. Normal hematological functions: neutrophils ≥ 1.5 x 109 cells/L, platelets ≥ 100 x 109 cells/L and Hb ≥ 10.0 g/dL).
16. Normal liver function: bilirubin < 1.5 x upper limit of the normal range (ULN), alkaline phosphatase and transaminases (ASAT, ALAT) < 3 x ULN.
17. Normal renal function: calculated (Cockcroft-Gault) or measured creatinine clearance ≥ 60 mL/min.
18. Absence of pregnancy:

    * Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and 6 months beyond stop of treatment and must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of investigational product;
    * Post menopause is defined as a documented serum follicle stimulating hormone (FSH) level ≥ 35 mIU/mL.
19. Females should not be breast feeding.
20. Patients must use a barrier method of contraception (e.g. condom for either male, female patients or partners of female patients) during TG6002 treatment period and for a minimum of 6 months following the last treatment with TG6002. In addition, to minimize the risk of pregnancy, female patients or female partners of male patients who are of childbearing potential must use an additional effective method of contraception (e.g. one of the following: hormonal contraception, occlusive cap, intrauterine device -IUD- or intrauterine system -IUS-, male sterilization, or true abstinence).
21. Before patient inclusion and study related procedures (that would not have been performed as part as standard care), written informed consent must be given according to International Conference on Harmonization-Good Clinical Practices (ICH/GCP), and national/local regulations.
22. Patient affiliated to social security. 23. Approval of participation, following discussion with the multidisciplinary board of neuro-oncology, in the best interest of patient and in absence of any other reasonable therapeutic alternative.

Exclusion Criteria:

1. Immunodeficiency:

   * CD4+ lymphocyte count <200/µL, in any case ;
   * HIV infection;
   * Immunosuppressive therapy, including high dose corticosteroids (at a dose ≥ 20 mg per day of prednisone or equivalent, at the inclusion visit).
2. History of severe exfoliative skin condition (e.g. eczema or atopic dermatitis) requiring systemic therapy for more than 4 weeks within 2 years of TG6002 treatment initiation.
3. History of a severe systemic reaction or side-effect as a result of a previous smallpox vaccination, such as systemic vaccinia, eczema vaccinatum, encephalitis, myocarditis, or pericarditis.
4. Patients with significant gastro-intestinal (GI) tract disease or resection leading to significant impairment of GI absorption or bacterial overgrowth.
5. Known deficiency in dihydropyrimidine dehydrogenase (DPD).
6. Hypersensitivity to flucytosine.
7. Hypersensitivity to egg proteins.
8. Hypersensitivity to gentamicin.
9. History of severe drug allergy.
10. Received systemic anti-cancer therapy within 4 weeks prior to first administration of TG6002.
11. Prior gene therapy.
12. Other medical condition or laboratory abnormality or active infection that in the judgment of the principal investigator may increase the risk associated with study participation or may interfere with interpretation of study results and /or otherwise make the patient inappropriate for entry into this study.
13. Patient unable or unwilling to comply with the protocol requirements and/or unwilling to sign an informed consent form.
14. Patient deprived of liberty or under legal protection measure.
15. Weight > 100kg.
16. Antiviral therapy (as ribavirin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participant with Dose Limiting Toxicities defined as Any of the following treatment-related adverse events (AEs) is evaluated and reported from Day 1 through Day 26; as assessed by NCI-CTCAE, version 4.03 | Through day 1 to day 26
  For Phase 1
  Assessment of safety and tolerability :
  Number of Participant with Dose Limiting Toxicities defined as Any of the following treatment-related adverse events (AEs) is evaluated and reported from Day 1 through Day 26; as assessed by NCI-CTCAE, version 4.03:
  * Any Grade 4 toxicity (except isolated Grade 4 lymphopenia lasting ≤ 7 days);
  * Grade 3 or 4 hypotension, disseminated intravascular coagulation (DIC), or allergic reaction/hypersensitivity;
  * Grade 3 skin lesions: ulcerative dermatitis or skin changes with pain interfering with function;
  * Number of skin lesions ≥ 10 corresponding to infection possibly or probably related to the administration of TG6002;
  * Grade 3 non-hematologic toxicity persisting for >7 days except increase in ASAT and/or ALAT (> 5x ULN), which may last >7 days if total bilirubin is normal or Grade 1;
  * Flu-like symptoms that do not respond to standard treatments;
  * Grade 3 hematologic toxicity persisting for > 7 days
Number of patients without documented tumor progression at 6 months from date of first TG6002 infusion according to Response Assessment Neuro-Oncology Criteria (Wen et al., 2010, JCO, PMID:20231676) | at 6 months according to RANO criteria
  For Phase 2a Number of patients without documented tumor progression at 6 months from date of first TG6002 infusion according to Response Assessment Neuro-Oncology Criteria (Wen et al., 2010, JCO, PMID:20231676)

SECONDARY OUTCOMES:
TG6002 recommended dose prior to the Phase 2a part of the study (RP2D) in combination with 5-FC (Maximum Plasma Concentration [Cmax]) | through study completion an average of 24 months
  Phase 1 The Recommended Phase 2 Dose (RP2D) is the dose recommended by the DSMB for Phase 2a investigation: the DSMB performed a complete review of the available results about safety and efficacy from the first phase
Overall Survival (OS) | through study completion : every 2 months the first year and then every 3 months from day 67 until the date of first documented progression or date of death from any cause wichever came first, assessed up to 51 months
  After the end of the treatment patients will be followed in the neurology department according to standards of care. In case of withdrawal, patients and/or their specified contacts could be contacted for survival and information on possible subsequent anti-cancer therapy and their general safety and efficacy
Relative quantification of circulating viral DNA | Day1, Day2, Day 15, Day 26
  Relative quantification of circulating viral DNA : Quantification of the viral genome by Quantitative Polymerase Chain Reaction
Blood pharmacokinetics of 5-FC | Day0, Day7, Day 14, Day 26
  Measurement of Cmax
Blood pharmacokinetics of 5-FC | Day0, Day7, Day 14, Day 26
  Measurement of Tmax
Blood pharmacokinetics of 5-FC | Day0, Day7, Day 14, Day 26
  Measurement of AUC
Blood pharmacokinetics of 5-FC | Day0, Day7, Day 14, Day 26
  Measurement of CI
Blood pharmacokinetics of 5-FC | Day0, Day7, Day 14, Day 26
  Measurement of MRT
Blood pharmacokinetics of 5-FC | Day0, Day7, Day 14, Day 26
  Measurement of Vd/F
Blood pharmacokinetics of 5-Fluorouraril (5-FU) | Day0, Day7, Day 14, Day 26
  Measurement of Cmax
Blood pharmacokinetics of 5-Fluorouraril (5-FU) | Day0, Day7, Day 14, Day 26
  Measurement of Tmax
Blood pharmacokinetics of 5-Fluorouraril (5-FU) | Day0, Day7, Day 14, Day 26
  Measurement of AUC
Blood pharmacokinetics of 5-Fluorouraril (5-FU) | Day0, Day7, Day 14, Day 26
  Measurement of CI
Blood pharmacokinetics of 5-Fluorouraril (5-FU) | Day0, Day7, Day 14, Day 26
  Measurement of MRT
Blood pharmacokinetics of 5-Fluorouraril (5-FU) | Day0, Day7, Day 14, Day 26
  Measurement of Vd/F
Blood pharmacokinetics of final metabolite a-fluoro-B-alanine(FBAL) | Day0, Day7, Day 14, Day 26
  Measurement of Cmax
Blood pharmacokinetics of final metabolite a-fluoro-B-alanine(FBAL) | Day0, Day7, Day 14, Day 26
  Measurement of AUC
Blood pharmacokinetics of final metabolite a-fluoro-B-alanine(FBAL) | Day0, Day7, Day 14, Day 26
  Measurement of Tmax
Blood pharmacokinetics of final metabolite a-fluoro-B-alanine(FBAL) | Day0, Day7, Day 14, Day 26
  Measurement of CI
Blood pharmacokinetics of final metabolite a-fluoro-B-alanine(FBAL) | Day0, Day7, Day 14, Day 26
  Measurement of MRT
Blood pharmacokinetics of final metabolite a-fluoro-B-alanine(FBAL) | Day0, Day7, Day 14, Day 26
  Measurement of Vd/F
Viral shedding in saliva, urine and feces | Day2, Day7
  by Quantitative Polymerase Chain Reaction and plaque assays (if q-PCR positive)
Humoral response | Baseline, Day 39
  Measurement of Blood anti-vaccinia virus and anti-FCU1 antibodies in blood
Isolation of peripheral blood mononuclear cells (PBMC); | Day 0, Day 26, Day 39
  Determine immunoprofile, potential predictive marker of efficacy
Metabolic Response | Baseline, Day 39, Day 67
  using PET-MRI ([18F]FDOPA -PET scans)
Safety and tolerability : Incidence of Treatment; evaluation of treatement-releated adverse events | through study completion an average of 51 months
  Complete review of serious and unserious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed IDBAIH, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided